CLINICAL TRIAL: NCT03723031
Title: The Efficacy and Safety of Intrauterine Misoprostol Versus Rectal Misoprostol in Reducing Blood Loss During and After Cesarean Section
Brief Title: Intrauterine Misoprostol Versus Rectal Misoprostol in Reducing Blood Loss During Cesarean Section
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1121980
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hemorrhage, Postpartum
Keywords: hemorrhage; misopristol; Cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rectal misopristol (Active Comparator): will receive 400 microgram misoprostol rectally preoperatively with urinary catheter insertion.
  Interventions: Drug: Misoprostol
- intrauterine misopristol (Active Comparator): will receive 400 microgram misoprostol inserted intrauterine (200 microgram at each cornu) intraoperatively following the delivery of the placenta.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 microgram (2 tablets) misoprostol ( cytotec, Pfizer, G.D. Searle LLC) inserted rectally (before CS) in rectal group or intrauterine (200 microgram at each cornu) intraoperatively following the delivery of the placenta in intrauterine group.
  Other Names: cytotec

SUMMARY:
98 pregnant women attending for CS will be randomized into 2 groups. Rectal misopristol group who will receive 400 microgram misoprostol rectally preoperatively with urinary catheter insertion and intrauterine misopristol group will receive 400 microgram misoprostol intrauterine (200 microgram at each cornu) intraoperatively following the delivery of the placenta. The estimated blood loss for each patient will be measured and data of both groups will be compared.

DETAILED DESCRIPTION:
The study we will include (98) pregnant women attending for cesarean delivery in the Kasr Elaini hospital (faculty of medicine - Cairo university).After signing informed written consent, all participants will be subjected to: Full medical history(including full obstetric history and current pregnancy history and the 1st day of last menstrual period), thorough clinical examination (general and full obstetric examination), obstetric ultrasonography (to confirm gestational age and the eligibility of the current pregnancy to participate in the study) and preoperative laboratory tests (including prothrombin time, prothrombin concentration, complete blood count, and liver and kidney function tests).

Group allocation: On the day of the cesarean delivery, participants will be randomly assigned in a 1:1 ratio into two groups; group A (Rectal misoprostol) and group B (Intrauterine misoprostol). Randomization will be performed using computer-generated random numbers and only the participants will be masked to the group allocation.

Group A (Rectal misoprostol - n=49) will receive 400 microgram misoprostol rectally preoperatively with urinary catheter insertion while group B (Intrauterine misoprostol n=49) will receive 400 microgram misoprostol (cytotec, Pfizer, G.D. Searle LLC) inserted intrauterine (200 microgram at each cornu) intraoperatively following the delivery of the placenta.

Following the delivery of the baby, patients in both groups will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h).

All cesarean sections will be done under spinal anesthesia by the following operative steps: pfannenstiel incision, transverse lower uterine segment incision, immediate cord clamping (< 30 seconds) and the placenta will be removed by controlled cord traction after its spontaneous separation, closure of uterus in 2 layers, closure of anterior abdominal wall in anatomical manner (adequate hemostasis will be ensured in all operative steps).

The number and the difference of weight of operative towels (before and after CS) and amount of blood in suction unit will be recorded.

The estimated blood loss for each patient will be measured and data of both groups will be compared.

In group A, the time interval between rectal misoprostol insertion and fetal delivery will be recorded together with the neonatal outcome (APGAR at 1 and 5 minutes, NICU admission and neonatal death).

Fluid monitoring will be performed through rate of infusion and urine output. A complete blood count test will be performed 12 hours after delivery.

All patients will be followed up for 24 hours following the delivery as regard occurrence of primary postpartum hemorrhage, the need for blood transfusion, misoprostol-related side effects in the first 6 hours (i.e. shivering, pyrexia more than 38 degree Centigrate, headache, nausea, vomiting with or without the need for anti-emetic drugs).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women candidate for CS.
* Full term singleton living pregnancies (> 37 weeks confirmed by the 1st day of the LMP or 1st trimesteric ultrasound scan).
* Spinal or epidural anesthesia for the CS.

Exclusion Criteria:

* Maternal Anemia (hemoglobin <9 g%)
* Maternal medical disorders (e.g. cardiac, renal, and hepatic diseases, or coagulopathies).
* Fetal anomalies or IUGR (estimated fetal weight below the 5th centile)
* Risk of obstetric hemorrhage (e.g. peripartum hemorrhage, abnormal placentation, previous history of uterine atony or postpartum hemorrhage).
* Women attending for emergency CS.
* More than 2 previous CS procedures.
* Prolonged procedure (more than 2 hours from skin incision to skin closure).
* History of prostaglandin allergy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
estimated blood loss during and after CS | within 12 hours after delivery
  EBL= EBV x { (Preoperative hematocrit - Postoperative hematocrit) ÷ Postoperative hematocrit} Where EBV is estimated blood volume of the patient in mL (equals weight in kg × 85).

SECONDARY OUTCOMES:
estimated blood loss during CS | within the CS procedure
  The number of operative towels used - The difference of weight of operative towels (before and after cs) plus the amount of blood in suction unit (we will calculate 1 gram of weight difference equal to 1 ml blood loss).
Use of additional ecbolics denoting uterine atony | within CS procedure
  additional 5 IU intravenous bolus oxytocin and 1mL [0.2 mg] intramuscular ergometrine with or without 600 microgram rectal misoprostol postoperatively)
The occurrence of any maternal side effects (in both groups) | within 24 hours after the CS procedure
  shivering, pyrexia >38C0, headache, nausea, vomiting with or without the need for antiemetic drugs
The occurrence of any fetal side effects (rectal group only) | within 24 hours after the CS procedure
  APGAR at 1 and 5 minutes, NICU admission and neonatal death

CONTACTS AND LOCATIONS:
Overall Officials: moutaz elsherbini, MD, Principal Investigator — Assistant professor of obstetrics and gynecology
Locations (1):
- Faculty of medicine - Cairo university, Cairo, Egypt

REFERENCES:
- [Derived] El-Sherbini MM, Maged AM, Helal OM, Awad MO, El-Attar SA, Sadek JA, ElKomy R, Dawoud MA. A comparative study between preoperative rectal misoprostol and intraoperative intrauterine administration in the reduction of blood loss during and after cesarean delivery: A randomized controlled trial. Int J Gynaecol Obstet. 2021 Apr;153(1):113-118. doi: 10.1002/ijgo.13426. Epub 2020 Nov 6. PMID 33064852